CLINICAL TRIAL: NCT00594490
Title: Adjunct Study for Silicone Gel-Filled Mammary Prosthesis
Brief Title: Evaluating the Effectiveness and Outcomes of Silicone Breast Prosthetics
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Mentor Worldwide, LLC (Industry)
Responsible Party: Principal Investigator, Gregory R. Evans, Professor, University of California, Irvine
Other Study IDs: 2001-2192
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: Breast, reconstruction, silicone
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Silicone: patients undergoing placement of silicone breast prosthetics

SUMMARY:
This trial will evaluate the outcome of placement of silicone breast prosthetics.

DETAILED DESCRIPTION:
Patients will be evaluated for complications following placement of silicone breast prostheses.

ELIGIBILITY:
Inclusion Criteria:

* over 18 undergoing breast reconstruction

Exclusion Criteria:

* patients with collagen vascular diseases, rheumatoid arthritis, scleroderma, etc.

Study Closed

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women undergoing breast reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2002-05-24 (Actual); Primary Completion 2013-12-19 (Actual); Study Completion 2013-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Evans, Principal Investigator — The University of California, Irvine
Locations (1):
- The University of California, Irvine, Orange, California, United States